CLINICAL TRIAL: NCT00745550
Title: A Phase 1/2 Study of Oral SB1518 in Subjects With Chronic Idiopathic Myelofibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: S*BIO (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SB1518-2008-003
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Myelofibrosis; Myeloproliferative Disorders; Polycythemia Vera; Essential Thrombocythemia
Keywords: SB1518; Chronic Idiopathic Myelofibrosis; Myeloproliferative disorders; Polycythemia Vera; Essential Thrombocythemia; JAK2 inhibitor
MeSH Terms: conditions — Primary Myelofibrosis; Myeloproliferative Disorders; Polycythemia Vera; Thrombocythemia, Essential | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SB1518 — SB1518 taken orally daily for 28 consecutive days in a 28-day cycle

SUMMARY:
The study consists of two phases: The first portion of the study is a Phase 1 dose escalation study to determine the maximum tolerated dose and the dose limiting toxicities of SB1518 when given as a single agent orally once daily in subjects with Chronic Idiopathic Myelofibrosis (CIMF) regardless of their JAK2 mutational status. The second portion of the study is a Phase 2 study to define the efficacy and safety profile of single agent SB1518 at the recommended dose in subjects with CIMF.

ELIGIBILITY:
Inclusion Criteria

* Subjects with CIMF (including post ET/PV MF) requiring therapy, including:
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Men of reproductive potential who can agree to practice effective contraception during the entire study period and for one month after the last study treatment
* Women of child-bearing potential who have a negative pregnancy test within 14 days prior to the first dose of study drug and can agree to practice effective contraception during the entire study period and for one month after the last study treatment, unless documentation of infertility exists
* Subjects who are able to understand and willing to sign the informed consent form

Exclusion Criteria

* Subjects with uncontrolled inter-current illness including, but not limited to, ongoing active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements as judged by treating physician. Subjects receiving antibiotics for infections that are under control may be included in the study unless the antibiotic is a CYP3A4 inducer/inhibitor
* Subjects known to be HIV-positive
* Subjects with known active hepatitis A, B, or C, or latent hepatitis B
* Women who are pregnant or lactating
* Subjects with prior radiation therapy to more than 20% of the hematopoietic marrow (prior radiation to spleen is allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Phase 1: to establish the maximum tolerated dose of SB1518 as a single agent when administered orally daily | Throughout the study
Phase 2: to assess the clinical benefit rate in subjects with CIMF who are treated with SB1518 at the recommended dose | Throughout the study

SECONDARY OUTCOMES:
Assess the safety and tolerability of SB1518, administered orally once daily in subjects with CIMF | Throughout the study
Assess the pharmacokinetic profile of SB1518 | Throughout the study
Assess the pharmacodynamic profile of SB1518 | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: John Seymour, M.D., Principal Investigator — Peter MacCallum Cancer Centre, Australia; Andrew Roberts, M.D., Principal Investigator — Melbourne Health; Bik To, MD, Principal Investigator — Royal Adelaide Hospital; Rami Komrokji, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute; Martha Wadleigh, MD, Principal Investigator — Dana-Farber Cancer Institute; Ruben Mesa, MD, Principal Investigator — Mayo Clinic
Locations (6):
- United States (3):
  - Mayo Clinic, Scottsdale, Arizona
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
- Australia (3):
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Royal Adelaide Hospital, Adelaide

REFERENCES:
- [Derived] Komrokji RS, Seymour JF, Roberts AW, Wadleigh M, To LB, Scherber R, Turba E, Dorr A, Zhu J, Wang L, Granston T, Campbell MS, Mesa RA. Results of a phase 2 study of pacritinib (SB1518), a JAK2/JAK2(V617F) inhibitor, in patients with myelofibrosis. Blood. 2015 Apr 23;125(17):2649-55. doi: 10.1182/blood-2013-02-484832. Epub 2015 Mar 11. PMID 25762180